CLINICAL TRIAL: NCT03238092
Title: Comparison Between Testosterone and Estradiol Over the Homogenization of Follicular Cohort: a Randomized Clinical Trial
Brief Title: Comparison Between Testosterone and Estradiol Over the Homogenization of Follicular Cohort
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hospital de Clinicas de Porto Alegre (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 67491417800005327
Record Dates: First submitted 2017-08-01; First posted 2017-08-03 (Actual); Last update posted 2017-08-03 (Actual); Status verified 2017-08

CONDITIONS: Fertility Disorders
Keywords: in vitro fertilization; estradiol; gnrh antagonist; testosterone
MeSH Terms: interventions — Testosterone; Estradiol

STUDY DESIGN:
Intervention Model Description: As a pre-treatment for in vitro fertilization, one arm will receive transdermic testosterone , one arm will receive oral estradiol and a third arm will be the control group, without pre-treatment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Estradiol group (Active Comparator): In the late luteal phase, the participant will receive estradiol 2mg and will take orally a total of 4mg per day (2mg in the morning and 2 mg in the night) until the next menstrual bleeding. After that, the patient will descontinue the medication and proceed to the regular in vitro fertilization protocol.
  Interventions: Drug: Estradiol
- Control group (No Intervention): No pre-treatment will be administrated. The regular in vitro fertilization protocol will be performed.
- Testosterone group (Experimental): Testosterone 25mg (10mg/g) transdermal during the late luteal phase, until the next menstrual bleeding.
  Interventions: Drug: Testosterone

INTERVENTIONS:
Drug: Testosterone — testosterone gel daily during the late luteal phase.
  Other Names: androgel
  Arms: Testosterone group
Drug: Estradiol — oral estradiol during the late luteal phase.
  Other Names: estradiol valerato
  Arms: Estradiol group

SUMMARY:
In vitro fertilization(IVF) with Gonadotropin-releasing hormone (GnRH) antagonist is one of the most used protocol for the treatment of infertile couples nowadays. Despite several advantages over GnRH agonist, the antagonist may be associated with a slightly reduction in pregnancy rates.

Several medications have been tested in order to increase ovarian response to ovulation induction, including estradiol and testosterone. A clinical trial in women with IVF indication will be performed and this women will be randomly assigned to receive topic testosterone, oral estradiol or no pre-treatment prior to IVF with human Chorionic Gonadotropin (hMG) and GnRH antagonist. The primary endpoint will be the size and number of follicles on the beginning of the cycle, after pre-treatment.

DETAILED DESCRIPTION:
One of the key-words to a successful IVF it is the response to the ovarian controlled stimulation. Nowadays, one of the most common protocols includes exogenous gonadotropins and GnRH antagonist, followed by IVF. The GnRH antagonist avoids the premature peak of LH and has advantages in relation to the GnRH agonist; however it might have a negative effect over the pregnancy rate. One possible explanation is the heterogeneity of the follicular cohort at the moment of ovarian puncture, due to the rise of FSH at luteal-follicular transition. The estrogen can inhibits this rise of Follicle-Stimulating Hormone (FSH), resulting in a more synchronic cohort. Previous studies have demonstrated a reduction in the cancellation rates with estradiol in the luteal phase of the cycle prior to the beginning of IVF using GnRH antagonist protocol, with a trend towards better quality of transferred embryos and better implantation rates when compared to the standard protocol with antagonist. The use of androgens is based on the assumption that they generate an increase in FSH receptors in the granulosa cells, increase in follicular growth and estrogen production, according to animal and human studies. Despite promising initial results, further studies are needed to evaluate the benefit of testosterone as a pretreatment in women undergoing IVF.

The study protocol is the following: Around the 20th day of the cycle prior to the choice of IVF, transvaginal pelvic ultrasound and serum progesterone dosage will be performed in all patients. After confirmation of ovulation and no contraindications for the continuation of the study, according to the randomization, testosterone gel, estradiol oral or no treatment will be initiated. Both medications will be continued until the first day of subsequent menstruation. After the menses, between the second and third day of the cycle, a new transvaginal ultrasound will be performed and blood tests will be collected for the dosage of FSH, Luteinizing Hormone (LH), progesterone and estradiol. On the same day, subcutaneous hMG (Menopur®) will be started at a dose between 150 and 300 IU / day, according to age and HAM, which will be subsequently adjusted according to the ovarian response on serial ultrasonography. When the largest follicle reaches a mean diameter of 14 mm, the GnRH antagonist (Orgalutran ®) will be initiated to prevent early LH peak, and monitored follicular growth with echography every 1-2 days. HCG will be administered at a dose of 10,000 IU (Choriomon®) when three or more follicles reach a mean diameter of 17 mm. After 36h, follicular puncture will be performed transvaginally, under general anesthesia. Embryo transfer will occur between the third and fifth day after in vitro fertilization. Luteal support will be given with administration of progesterone 600 mg / day vaginally, initiated after the transfer and maintained until the first trimester of pregnancy if it occurs. Serum beta-HCG measurement will be performed on the 12th day after transfer, for evaluation of pregnancy implantation. Clinical gestation will be considered when there is evidence of intrauterine embryo with cardiac beats present on the ultrasound, after 6 weeks of transfer of the embryo (s).

ELIGIBILITY:
Inclusion Criteria:

* Regular cycles (between 25-34 days)
* In vitro fertilization indication for male cause, unexplained infertility or tubal factor
* Both ovaries
* Thyroid-stimulating hormone(TSH) < 2,5 mU/L
* Anti-Müllerian hormone (AMH) between 1-5 ng/ml
* Body Mass Index (BMI) < 30

Exclusion Criteria:

* Ovarian surgery
* Endometriosis
* Endocrinology or metabolic disorder
* Polycystic ovary syndrome (PCOS)
* Poor Ovarian Response (according to Bologna criteria)

Ages: 18 Years to 39 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 26 (Estimated)
Dates: Start 2017-08 (Estimated); Primary Completion 2018-01 (Estimated); Study Completion 2018-03 (Estimated)

PRIMARY OUTCOMES:
number of antral follicles | 15 days after intervention
  Number of follicles measured by transvaginal ultrasound during the first or second day after menstruation

SECONDARY OUTCOMES:
follicular cohort homogeneity | 15 days after intervention
  The comparison of medium follicular diameter (also measured by transvaginal ultrasound) of all the follicles during the first or second day after menstruation
metaphase II oocytes | 30 days
  the number of metaphase II oocytes
gonadotrophin use | 30 days
  number of units of gonadotrophin used during the in vitro fertilization protocol
number of embryos | 30 days
  the number of embryos assessed during the in vitro fertilization
pregnancy | 6 weeks
  clinical pregnancy, defined by the evidence of intrauterine embryo in the ultrasound

CONTACTS AND LOCATIONS:
Overall Officials: João Sabino, PhD, Principal Investigator — Hospital de Clinicas de Porto Alegre

IPD SHARING:
Plan to Share IPD: Undecided